CLINICAL TRIAL: NCT01962116
Title: Citrate Versus Heparin for the Lock of Non-tunneled Hemodialysis Catheters in Patients Hospitalised in ICU = Multicentre, Controlled, Randomised Superiority Trial
Brief Title: Citrate Versus Heparin for the Lock of Non-tunneled Hemodialysis Catheters in Patients Hospitalised in ICU
Acronym: VERROU-REA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QUENOT DB 2012
Record Dates: First submitted 2013-08-27; First posted 2013-10-14 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Patients With Acute Renal Insufficiency
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin lock (Placebo Comparator)
  Interventions: Drug: unfractionated heparin
- Citrate lock (Experimental)
  Interventions: Drug: Citrate 4%

INTERVENTIONS:
Drug: Citrate 4%
  Arms: Citrate lock
Drug: unfractionated heparin
  Arms: Heparin lock

SUMMARY:
After obtaining written informed consent and inclusion, patients will be randomised into 2 groups for the type of dialysis catheter lock:

* The first group will have a citrate lock
* The second group will have a heparin lock Patients will be stratified according to the centre and type of Renal Replacement Therapy (RRT) continuous or intermittent.

The daily surveillance of patients will not be different from the usual surveillance of patients on Renal Replacement Therapy.

The hemodialysis catheters used will be specific Renal Replacement Therapy catheters.

The decision to withdraw the catheter will be made by the investigator and based on clinical criteria (complications related to the catheter, termination of Renal Replacement Therapy…)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Requiring RRT for acute renal insufficiency
* For which a 1st non-tunneled catheter is placed
* In the jugular or femoral position
* After written informed consent has been obtained from the patient, a member of the family or a person of trust

Exclusion Criteria:

* Patient presenting active poorly controlled bleeding
* Known allergy to citrate
* Acute liver failure (Prothrombin level <30%)
* Thrombopenia < 30 000/mm3
* Known or suspected heparin-induced thrombopenia
* Known systemic bacterial infection at the time the catheter is placed
* catheter in the subclavicular position
* Persons not affiliated to a national health insurance scheme
* Pregnant women
* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of event-free survival of the first non-tunneled hemodialysis catheter (defined at the time in days from catheter insertion to withdrawal whatever the reason) | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France

REFERENCES:
- [Result] Quenot JP, Helms J, Bourredjem A, Dargent A, Meziani F, Badie J, Blasco G, Piton G, Capellier G, Mezher C, Rebibou JM, Nadji A, Crepin T, Barbar SD, Fleck C, Cransac A, Boulin M, Binquet C, Soudry-Faure A, Bruyere R; VERROU-REA Trial Investigators and the CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). Trisodium citrate 4% versus heparin as a catheter lock for non-tunneled hemodialysis catheters in critically ill patients: a multicenter, randomized clinical trial. Ann Intensive Care. 2019 Jul 1;9(1):75. doi: 10.1186/s13613-019-0553-4. PMID 31264073
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Bruyere R, Soudry-Faure A, Capellier G, Binquet C, Nadji A, Torner S, Blasco G, Yannaraki M, Barbar SD, Quenot JP. Comparison of heparin to citrate as a catheter locking solution for non-tunneled central venous hemodialysis catheters in patients requiring renal replacement therapy for acute renal failure (VERROU-REA study): study protocol for a randomized controlled trial. Trials. 2014 Nov 19;15:449. doi: 10.1186/1745-6215-15-449. PMID 25409678